CLINICAL TRIAL: NCT03726788
Title: Analysis of Antalgic Efficacy of an Intra Articular Injection of Botulinum Toxin Versus Corticoids in Gonarthrosis by Perfusion MRI:a Superiority, Randomized, Controlled, Double Blind Study
Brief Title: Intra Articular Injection of Botulinum Toxin Versus Corticoids in Gonarthrosis
Acronym: TOXART
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: discontinuation of the study
Sponsor: Lille Catholic University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC-P0037
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Joint Diseases; Knee; Therapeutics; Magnetic Resonance Imaging
Keywords: knee; Arthrosis; Botulinum toxin; Magnetic Resonance Imaging
MeSH Terms: conditions — Joint Diseases; Osteoarthritis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only pharmacists and radiologists know the patient's randomizing arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botulinum Toxin Type A 100U (Experimental): one intra-articular injection in the painful knee 30 days after the inclusion visit
  Interventions: Drug: Botulinum Toxin Type A 100U
- Botulinum Toxin Type A 200U (Experimental): one intra-articular injection in the painful knee 30 days after the inclusion visit
  Interventions: Drug: Botulinum Toxin Type A 200U
- Triamcinolone Hexacetonide 20 MG/ML (Active Comparator): one intra-articular injection in the painful knee 30 days after the inclusion visit
  Interventions: Drug: Triamcinolone Hexacetonide Inj Susp 20 MG/ML

INTERVENTIONS:
Drug: Botulinum Toxin Type A 100U — one intra-articular injection of 100 U of botulinum toxin type A, diluted in 2 ml of 0.9% SSI
  Other Names: Botox 100 UNT Injection
  Arms: Botulinum Toxin Type A 100U
Drug: Botulinum Toxin Type A 200U — one intra-articular injection of 200 U of botulinum toxin type A, diluted in 4 ml of 0.9% SSI
  Other Names: Botox 200 UNT Injection
  Arms: Botulinum Toxin Type A 200U
Drug: Triamcinolone Hexacetonide Inj Susp 20 MG/ML — one intra-articular injection of 2 ml Triamcinolone Hexacetonide
  Other Names: HEXATRIONE
  Arms: Triamcinolone Hexacetonide 20 MG/ML

SUMMARY:
We believe we can demonstrate a link between the analgesic action of intra-articular injection of botulinum toxin and synovial inflammation by Dynamic Contrast Enhancement (DCE) perfusion Magnetic Resonance Imaging (MRI).

DETAILED DESCRIPTION:
Knee osteoarthritis is one of the most common causes of joint pain and functional disability in the general population.

Intra-articular infiltrations of corticoids are indicated for painful crisis especially if accompanied of effusion. However, this effect lasts only 2 weeks.

Given the lack of effective long-term medical-infiltrative treatment, we believe that botulinum toxin type A could be used by its direct action on mediators of neuro-gene inflammation at the joint level and its indirect medullary action by retrograde migration.

To date, 2 published randomized controlled trials and one unpublished Phase Ib clinical trial have shown that botulinum toxin injected intraarticularly improves pain and functionality in gonarthrosis.

Dynamic Contrast Enhancement (DCE) Magnetic Resonance Imaging (MRI) demonstrated the correlation between synovial inflammation and pain in gonarthrosis in a cohort of 454 subjects. It has also made it possible, via the monitoring of synovial inflammation, to demonstrate the efficacy of treatments in patients suffering from rheumatoid arthritis in the early phase, juvenile chronic arthritis or osteoarthritis.

DCE MRI perfusion therefore appears here as the technique of choice to follow the evolution of synovial inflammation after botulinum toxin injection in patients with symptomatic gonarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Presenting gonarthrosis of degenerative origin, Kellgren/Lawrence Radiological Stage I to III, with a maturity of more than 18 months
* With pain intensity greater than or equal to 50/100 on an VAS
* In case of bilateral gonarthrosis, the VAS of the contralateral knee must be less than or equal to 30/100
* Presenting a failure of conventional per os treatments (non-steroidal anti-inflammatory drugs, analgesics)
* Affiliated with a social security scheme
* For women of childbearing age:

  * effective contraception for the duration of the study

Exclusion Criteria:

* Patient presenting at the time of the inclusion visit: an inflammatory attack, septic or inflammatory arthritis, a generalized infectious episode in progress
* Local or regional local skin lesion
* Need of an arthroplasty within the next 12 months
* Having received corticosteroids or other molecules in intra-articular infiltration in the last 6 months
* History of traumatic knee injury (bone injury in the past 24 months), bone, ligament or meniscal surgery in the past 24 months
* History of disabling peripheral nerve injury
* Severe bleeding disorders, anticoagulant treatment in progress or double antiplatelet aggregation
* BMI > 35 kg/m2
* Coxarthrosis with projected knee pain
* Pregnant or breastfeeding woman
* Patient under guardianship and protection of justice
* Allergy/contraindication to botulinum toxin type A, corticoids
* Usual contraindication to MRI
* Allergy to the contrast product

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Assesment of vascularization by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) according to the % Area Under the Curve (AUC) of perfusion value | one month post-injection

SECONDARY OUTCOMES:
Pain analysis by the visual analogue scale (VAS) | during the first 3 months after injection
  Evolution kinetics of daily pain collected during the first 3 months post-injection allowing to deduce the onset and duration of analgesic efficacy in number of days. The pain VAS is a continuous scale comprised of a horizontal line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "pain as bad as it could be" (score of 100 [100-mm scale])
Joint amplitude measured by goniometry | at 1, 3, 6 month post-injection
  To measure range of motion of the knee
Western Ontario McMaster University Osteoarthritis (WOMAC) Index | at 1, 3, 6 month post-injection
  An arthritic pain scoring system ranging from 0-no pain/disability to 100-most severe pain/disability
Two minutes walk | at 1, 3, 6 month post-injection
  This test measure the distance walked in two minutes
Frequency of consumption of analgesics | at 1, 3, 6 month post-injection
Amount of consumption of analgesics | at 1, 3, 6 month post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Hichem Khenioui, MD, Principal Investigator — GHICL
Locations (1):
- Lille Catholic University, Lille, France

IPD SHARING:
Plan to Share IPD: No